CLINICAL TRIAL: NCT07078214
Title: The Effect of Backward Walking on Toe Walking Behaviors in a Child With Autism Spectrum Disorder: Single-participant (Subject) Experimental Research
Brief Title: Backward Walking Effects on Toe Walking in a Child With ASD: Single-Case Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Ekrem AKBUGA, PhD, Assistant Proffessor, Giresun University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRU-SBF-EA-001
Record Dates: First submitted 2025-06-28; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Toe Walking Behaviors; Backward Walking
Keywords: Autism; Backward walking; Toe walking
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Intervention Model Description: This study is a prospective research based on single-subject experimental design. Model A-B-A (Reversal Design) was preferred because it was desired that the provided benefit continue in favor of the child without interruption. In this design, the baseline level of the targeted behavior is determined, and during the implementation phase, the behavior is expected to gradually change toward the main goal, and the effects of the independent variable are monitored during a second baseline phase (withdrawal or monitoring). Additionally, the principles and instructions in the SCRIBE guidelines were taken into consideration in the design and implementation of this study. This guideline is a reporting manual for single-participant designs in behavioral interventions.
Masking Description: Blinding for the Participant: To obtain reliable data from gait measurements, the participant is asked to exhibit their natural gait on the walking platform. It was observed that the child exhibited natural gait because the participant did not focus much on environmental elements and did not realize that the participant was being subjected to measurement. This situation was considered as blinding for the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A child with ASD exhibiting TWB (pseudonym "Daisy") (Experimental): Intervention Type: Backward walking exercise (treadmill-based) Frequency: 5 days per week Duration: 9 weeks (intervention phase) Session duration: 10-12 minutes/session; 2 sessions Intensity: Adapted according to participant's developmental level and safety requirements Implementation setting: In a controlled laboratory environment, specially adapted treadmill Supervision: Continuous supervision by trained researchers Measurement: Plantar surface area measurement using pedobarographic analysis Safety protocol: Safety measures adapted to individual needs
  Interventions: Other: Foot Sole Surface Area Measurements; Other: Walking Exercise Program and Implementation Process

INTERVENTIONS:
Other: Foot Sole Surface Area Measurements — The child's TWB was measured using the BTS P-Walk platform [2440x740x8 mm, 12,000 sensors] with an additional 500mm sensor-free mat for accurate start/end measurements. The system focused on foot-ground contact surface area data.Before measurements, the child familiarized herself with the platform through play. All walks were barefoot, with at least 3 attempts per assessment and the clearest data selected. To encourage platform crossing, the child carried a small object to her mother waiting opposite. To prevent upper extremity interference with gait, only return walks (without object) were analyzed for measurement.
Other: Walking Exercise Program and Implementation Process — The backward walking exercise program was performed on a treadmill at 1±0.2 km/h speed, conducted 5 days per week between 14:00-15:00 hours when the child was most alert according to maternal reports. Initially planned for minimum 5-minute sessions with gradual increases, but the child's short attention span and unfamiliarity with backward walking limited sessions to 3 minutes during first two days. Favorite cartoons displayed via tablet during sessions successfully enabled gradual time increases. Week 1 progressed from 3-5 minutes daily. Weeks 2-5 showed progressive increases to 6-9 minutes with sessions increased to 2 daily, separated by 10-15 minute play breaks. From week 6 onwards, two 10±0.2 minute sessions continued daily. Starting week 3, sessions were restructured as 5 minutes backward + 1 minute forward + 2-7 minutes backward walking to combat attention deficits after 5 minutes, improving exercise efficiency.

SUMMARY:
This study tested the hypothesis that backward walking exercises can reduce Toe Walking Behaviors (TWB) in children with ASD and emphasized the importance of pedobarographic measurements for quantitative TWB assessment.

DETAILED DESCRIPTION:
Study Description: Backward Walking Exercise Intervention for Toe Walking in Children with Autism Spectrum Disorder Study Overview This research study investigates whether backward walking exercises can help reduce toe walking behavior in young children with Autism Spectrum Disorder (ASD). Toe walking is a common movement pattern where children walk on their toes instead of using their whole foot, which can affect balance, coordination, and overall development.

Background and Importance Children with Autism Spectrum Disorder often develop unusual walking patterns, including toe walking, which can impact their physical development and daily activities. Traditional approaches to address this behavior have shown limited success, making it important to explore new, evidence-based interventions that can be easily implemented and monitored.

Study Design and Approach

This study uses a single-subject research design, which allows for detailed examination of individual responses to treatment. The research follows a structured A-B-A pattern:

Baseline Phase (1 week): Researchers measure the child's natural walking pattern without any intervention Implementation Phase (9 weeks): The child participates in backward walking exercises on a treadmill Monitoring Phase (1 week): Researchers observe whether improvements continue after stopping the exercises Participants The study focuses on young children (approximately 3-4 years old) who have been diagnosed with Autism Spectrum Disorder and demonstrate persistent toe walking behavior. Participant is carefully selected to ensure they can safely participate in treadmill-based exercises.

What the Study Involves Exercise Program: Children participate in backward walking exercises on a specially adapted treadmill, designed to be safe and appropriate for their developmental level. These sessions occur 5 days per week during the treatment phase.

Measurement Technology: The study uses advanced foot pressure measurement technology (pedobarographic analysis) to precisely track how much of the child's foot touches the ground during walking. This provides objective, quantitative data about walking patterns.

Monitoring and Safety: All activities are supervised by trained researchers and adapted to each child's individual needs and abilities.

Study Duration

The complete study spans 11 weeks:

Week 1: Baseline measurements Weeks 2-10: Backward walking exercise intervention Week 11: Follow-up monitoring Potential Benefits This research may help establish backward walking exercises as an effective, non-invasive intervention for addressing toe walking in children with ASD. The findings could contribute to improved physical therapy approaches and better developmental outcomes for children with autism.

Scientific Significance This study employs rigorous single-subject methodology following established research guidelines (SCRIBE) to ensure reliable and valid results. The use of objective measurement technology provides precise data that can help clinicians and families make informed decisions about treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* It was required that the participant be diagnosed with ASD, exhibit TWB, be able to follow simple instructions, have no health problems other than ASD, and not have participated in any exercise program or physical therapy rehabilitation. It has been reported by orthopedic and physical therapy specialists, whom the parents had previously consulted, that the child exhibits TWB with ASD characteristics only, without any musculoskeletal problems.

Exclusion Criteria:

* Children with any musculoskeletal problems, diagnoses other than ASD (such as cerebral palsy, etc.), or those who had previously undergone surgical operations on the lower extremities were not included in the study.

Min Age: 3 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Foot Sole Surface Area Measurements | 11weeks (55 days)- 9 weeks of implementation
  Toe walking behavior (TWB) was measured using the BTS P-Walk platform [2440x740x8 mm with 2400x500 mm sensorized area containing 12,000 sensors]. A 500 mm sensor-free mat was added at platform ends for accurate start/end measurements. The system focused on foot-ground contact surface area data relevant to this study's objectives. Before measurements, the child familiarized herself with the platform through play activities to ensure comfort. All assessments were conducted barefoot with at least three walks per session, selecting the clearest data for analysis. To encourage natural platform crossing, the child carried a small object to her mother waiting opposite. To prevent upper extremity interference with gait patterns, only return walks without the object were analyzed, ensuring accurate toe walking measurements unaffected by carrying tasks or arm movements during the assessment protocol. Changes assessed using visual analysis and statistical measures including ES calculations.

CONTACTS AND LOCATIONS:
Locations (1):
- Giresun University, Sport Science Faculty, Güre Campus, Giresun, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not want to share my data. I am sorry.